CLINICAL TRIAL: NCT03050086
Title: An Open Label Phase 2 Feasibility Study to Assess the Safety and Efficacy of BPX-04 Minocycline Topical Gel in Treatment of Moderate to Severe Papulopustular Rosacea (BPX-01-C05)
Brief Title: Open Label Phase 2 Feasibility Study of BPX-04 Topical Minocycline Gel in Rosacea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioPharmX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPX-01-C05
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Moderate to Severe Papulopustular Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BPX-04 1% Minocycline Topical Gel (Experimental): once daily topical administration of 1% minocycline gel to the face
  Interventions: Drug: BPX-04 1% minocycline topical gel
- BPX-04 2% Minocycline Topical Gel (Experimental): once daily topical administration of 2% minocycline gel to the face
  Interventions: Drug: BPX-04 2% minocycline topical gel
- BPX-01 Vehicle Topical Gel (Placebo Comparator): once daily topical administration of vehicle gel to the face
  Interventions: Drug: BPX-04 vehicle topical gel

INTERVENTIONS:
Drug: BPX-04 1% minocycline topical gel — once daily administration of topical minocycline gel to face
  Arms: BPX-04 1% Minocycline Topical Gel
Drug: BPX-04 2% minocycline topical gel — once daily administration of topical minocycline gel to face
  Arms: BPX-04 2% Minocycline Topical Gel
Drug: BPX-04 vehicle topical gel — once daily administration of topical minocycline gel to face
  Arms: BPX-01 Vehicle Topical Gel

SUMMARY:
An open label feasibility study using BPX-04 topical minocycline gel in papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age at the time of consent.
2. Subjects do not have any medical conditions, other than rosacea, that in the opinion of the investigator, put the subject at unacceptable risk or could interfere with study assessments or integrity of the data.
3. A clinical diagnosis of moderate to severe (Grade 3 or 4) facial rosacea (papulopustular (Subtype 2) or mixed erythematotelangiectatic (Subtype 1) and papulopustular (Subtype 2)) as determined by the Investigator's Global Assessment (IGA) at Visit 1/Screening.
4. Female subjects of childbearing potential (including pre-puberty) are willing to use effective contraceptive method for at least 28 days before baseline (Day 0) and at least 28 days after the last study product administration or have a sterilized or same-sex partner for the duration of the study. Hormonal contraceptives must be on a stable dose for at least 12 weeks before baseline (Day 0). Subjects using low dose oral contraceptives must use a second form of birth control (e.g., barrier method such as condoms with spermicide).

   Note: Female subjects of non-childbearing potential are defined as follows:
   1. Female subjects who have had surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation);
   2. Female subjects who have had a cessation of menses for at least 12 months and a follicle-stimulating hormone (FSH) test confirming non-childbearing potential (refer to the central laboratory reference range for menopausal women) or cessation of menses for at least 24 months without FSH levels confirmed;
5. Female subjects of childbearing potential must have a negative urine pregnancy test at screening and baseline (Day 0).
6. Treatment with hormonal therapy must be on a stable dose and frequency for at least 12 weeks before baseline (Day 0) and must remain stable throughout the study.
7. Subjects who use make-up, facial moisturizers, creams, lotions, cleansers and/or sunscreens must have used the same product brands/types for a minimum period of 14 days prior to baseline (Day 0), must agree not to change brand/type or frequency of use throughout the study and must agree not to use make-up, facial moisturizers, creams, lotions, cleansers and/or sunscreens on the clinic visit days before the visit.
8. Subjects must be capable of giving informed consent and the written informed consent must be obtained prior to any study-related procedures.

Exclusion Criteria:

1. Have a history of skin disease, presence of skin condition or excessive facial hair the PI believes would interfere with the study
2. Have moderate or severe rhinophyma, severe telangiectasia or plaque-like facial edema
3. Have rosacea conglobata or fulminans, corticosteroid induced rosacea or facial erythrosis other than rosacea
4. Have ocular rosacea of a severity that requires systemic treatment
5. Have a history of any adverse reaction to minocycline or other tetracycline class antibiotic
6. Have a clinically significant chemistry or hematology value at baseline or have an ALT or AST at screening that is greater than or equal to 2x normal
7. Have conditions or factors that the PI believes may affect the response of the skin or the interpretation of the results
8. Participated in any clinical study with exposure to any investigational treatment or product within the previous 30 days, or plan on concurrent participation in other studies
9. Have used on the face an OTC topical medication for the treatment of rosacea within 4 weeks prior to baseline.
10. Have used prescription topical (on the face) or oral antibiotics or corticosteroids within 4 weeks prior to baseline.
11. Have had a facial procedure such as chemical peel, laser, microdermabrasion within 8 weeks prior to baseline
12. Have received photodynamic therapy or phototherapy with blue or red light within 12 weeks prior to baseline
13. Have used an oral retinoid within 6 months or a topical retinoid within 3 months prior to baseline
14. Current drug or alcohol abuse
15. Female subject who is breastfeeding, pregnant or who is planning a pregnancy during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment | 12 weeks
  papules, pustules and erythema

SECONDARY OUTCOMES:
Lesion count | 12 weeks
  papules and pustules

CONTACTS AND LOCATIONS:
Overall Officials: AnnaMarie Daniels, Study Director — BioPharmX, Inc.
Locations (1):
- Study Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No